CLINICAL TRIAL: NCT03735706
Title: The Relationship Between COntrast Media Volume and Tube voLtage in Computed Tomography of the Liver, for Optimal Enhancement Based on Total Body Weight: A Randomized Controlled Trial. [COMpLEx Trial]
Brief Title: Relationship Between Contrast Media Volume and Tube Voltage in CT for Optimal Liver Enhancement, Based on Body Weight.
Acronym: COMpLEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: NL66971.068.18
Record Dates: First submitted 2018-10-31; First posted 2018-11-08 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Radiation; Contrast Media; Liver; Body Weight
Keywords: Radiation; Contrast media; Liver; Body Weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Intervention Model Description: randomized controlled trial with 4 study arms.
Who Masked: Participant, Care Provider, Investigator
Masking Description: A computer random number generator prepares the randomization schedule in a 1:1:1:1 manner, which is balanced randomization. Stratification is performed, based on age (< 60 and ≥ 60 years) and weight < 75 and ≥ 75 kg). Variable block randomization will distribute patients equally over time.
  The blinding and randomization process will be conducted by Clinical Trial Centre Maastricht (CTCM, www.CTCM.nl) with a randomization program (ALEA) designed for usage of different techniques.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group - 120 kV - 0.521 g I/kg (Active Comparator): Weight is measured prior to the scan. Before performing the contrast enhanced CT scan(s), an unenhanced slice through the liver, at the level of the portal vein, is performed.
  Contrast media injection protocol with a standard dosing factor of 0.521 g I/kg of TBW and a tube voltage of 120 kV.
  The intervention is the application of a standard contrast media volume and a standard tube voltage of 120 kV.
  Interventions: Radiation: Unenhanced slice; Diagnostic Test: Weight
- 90 kV - 0.521 g I/kg (Experimental): Weight is measured prior to the scan. Before performing the contrast enhanced CT scan(s), an unenhanced slice through the liver, at the level of the portal vein, is performed.
  Contrast media injection protocol with a standard dosing factor of 0.521 g I/kg of TBW.
  A radiation dose reduction from 120 to 90 kV.
  The intervention is a change in tube voltage to 90 kV, compared to group 1. The other intervention; contrast media volume, is unchanged compared to group 1.
  Interventions: Radiation: Radiation dose reduction; Radiation: Unenhanced slice; Diagnostic Test: Weight
- 100 kV - 0.417 g I/kg (Experimental): Weight is measured prior to the scan. Before performing the contrast enhanced CT scan(s), an unenhanced slice through the liver, at the level of the portal vein, is performed.
  Contrast media volume reduction with a dosing factor of 0.417 g I/kg of TBW. A radiation dose reduction from 120 to 100 kV compared to group 1.
  The intervention is a change in tube voltage to 100 kV, compared to group 1. The other intervention is a change in contrast media volume, which is adapted to the tube voltage used and therefore lowered to 0.417 g I/kg.
  Interventions: Radiation: Radiation dose reduction; Other: Contrast media volume reduction; Radiation: Unenhanced slice; Diagnostic Test: Weight
- 90 kV - 0.365 g I/kg (Experimental): Weight is measured prior to the scan. Before performing the contrast enhanced CT scan(s), an unenhanced slice through the liver, at the level of the portal vein, is performed.
  Contrast media volume reduction with a dosing factor of 0.365 g I/kg of TBW. A radiation dose reduction from 120 to 90 kV compared to group 1.
  The intervention is a change in tube voltage to 90 kV, compared to group 1. The other intervention is a change in contrast media volume, which is adapted to the tube voltage used and therefore lowered to 0.365 g I/kg.
  Interventions: Radiation: Radiation dose reduction; Other: Contrast media volume reduction; Radiation: Unenhanced slice; Diagnostic Test: Weight

INTERVENTIONS:
Radiation: Radiation dose reduction — The radiation dose is is different between groups
  Arms: 100 kV - 0.417 g I/kg; 90 kV - 0.365 g I/kg; 90 kV - 0.521 g I/kg
Other: Contrast media volume reduction — Contrast media volume is different between groups
  Arms: 100 kV - 0.417 g I/kg; 90 kV - 0.365 g I/kg
Radiation: Unenhanced slice — One unenhanced slice at the level of the portal vein will be added to the protocol before administration of contrast media. It will only take a minute to perform this extra slice. The patient does not have to visit the department a second time and no (extra) contrast is needed for this slice.
Diagnostic Test: Weight — A weighing scale is used to measure a patients body weight right before the scan.

SUMMARY:
Computed Tomography (CT) is widely used in abdominal imaging for a variety of indications. Contrast media (CM) is used to enhance vascular structures and organ parenchyma. Attenuation of the liver makes it possible to recognize hypo- and hypervascular lesions, which are often invisible on unenhanced CT images. Lesions can only be detected in case they are large enough and the contrast with the background is high enough. Heiken et al. showed already in 1995 that a difference in Hounsfield Units (HU) of at least 50 HU is needed to be able to recognize liver lesions [1]. On the other hand, patients should not receive more CM than necessarily, because of possible underlying physiological effects [2-4]. Although there has been some controversy about this recently, there is no need to give patients more CM than needed, because of increased costs, no quality improvement and their might still be a relationship with contrast induced nephropathy (CIN) [5].

Recent publications suggested individualization of injection protocols that can be based on either total body weight (TBW) or lean body weight (LBW) [6-9]. In the investigators department an injection protocol based on TBW is currently used.

Besides the CM injection parameters, scanner parameters are of influence on the attenuation as well. Because of recent technical developments it became possible to reach a good image quality (IQ) at lower tube voltages [10]. When the x-ray output comes closer to the 33 keV k-edge of Iodine, attenuation increases. In short, decreasing the tube voltage increases the attenuation of iodine. Scanning at a lower tube voltage therefore gives rise to even lower CM volumes. Lastly, it would be revolutionary to accomplish a liver enhancement that is homogenous, sufficient for lesion detection and comparable between patients and in the same patients, regardless of weight and scanner settings used.

DETAILED DESCRIPTION:
Computed Tomography (CT) is a non-invasive imaging tool, used for a great variety of indications. Contrast media (CM) is used to enhance vascular structures and organ parenchyma. The visibility of liver lesions depends mainly on the ratio between the size and the difference of the lesion to the background. A large lesion might be visible without administration of CM, whilst a smaller lesion needs the addition of CM to become visible. Additionally, CM can be useful in the characterization of liver lesions. Heiken et al. (1995) found that an attenuation of the parenchyma after CM administration of at least ∆ 50 Hounsfield units (HU) compared to an unenhanced scan (in the same patient) is necessary to recognize liver lesions. This study proposed a dosing factor of 0.521 g I/kg to be necessary to reach such attenuation at a tube voltage of 120 kV [1].

The parenchymal enhancement depends on patient, CT scanner and CM factors. Weight, height, cardiac output, age, gender, venous access, breath-holding, renal function and comorbidity all fall under patient factors [8]. Recently much research showed preferable outcomes for individualized CM injection protocols, in which the contrast bolus is adapted to patient TBW, LBW or body surface area (BSA) [6, 7, 9, 13-15]. In a recent feasibility study in the department of the investigators, the attenuation of the liver parenchyma was evaluated. Results showed that a body weight adapted CM injection protocol resulted in more homogeneous liver enhancement compared to a fixed CM dose (not published yet).

With recent technological developments in X-ray tube technology it became possible to use lower tube voltages. As a result making it possible to perform scans with a sufficient image quality (IQ) and a low tube voltage and therefore a lower radiation dose [10]. Another advantage lies in the fact that reducing the tube voltage, approaching 33 keV k-edge of iodine, results in an increase in attenuation of the iodine. The new technological developments make it possible to reduce the radiation dose and CM volume at the same time. So reducing the tube voltage, makes it also possible to reduce the CM volume.

As recommended by the supplier, it is possible to calculate the total iodine load (TIL) that can be spared with the use of lower kV settings [16]. A reduction of 10 kV should result in a 10% reduction in CM volume. Reducing the tube voltage from 120 to 90 kV should therefore lead to a 30% reduction in CM volume. As mentioned before it is preferred to use an individualized CM injection protocol based on TBW or LBW. For this study, this theory is adapted to the concept of TBW. The following indicates which dosing factors should be used for each kV setting, based on the recommendations mentioned in the above.

120 kV -> 0.521 g I/kg 110 kV -> 0.469 g I/kg 100 kV -> 0.417 g I/kg 90 kV -> 0.365 g I/kg 80 kV -> 0.313 g I/kg 70 kV -> 0.261 g I/kg

The aim of present study is to investigate if adapting the dosing factor based on TBW and therefore the CM volume to the tube voltage used, results in a more homogeneous liver enhancement. The hypothesis is to find a more homogeneous enhancement between patients and in the same patient, regardless of body composition and tube voltage used.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for abdominal CT in portal venous phase
* Patients ≥ 18 years and competent to sign an informed consent

Exclusion Criteria:

* Hemodynamic instability
* Pregnancy
* Renal insufficiency (defined as Glomerular Filtration Rate (GFR) < 30 mL/min/1,73m2 [Odin protocol 004720])
* Iodine allergy (Odin protocol 022199)
* Age <18 years
* Absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
A liver attenuation (Δ HU) | Measurement for each scan is performed withing 1 month after the scan.
  The attenuation of the liver parenchyma as assessed by measuring the Hounsfield units (HU) of the liver parenchyma in an unenhanced CT scan and a scan in portal venous phase. The difference between the enhanced and unenhanced CT scan is the Δ HU. It is expected that scans in all groups have a Δ HU of at least 50 HU, which is considered sufficient. Therefore it is a non-inferiority outcome.

SECONDARY OUTCOMES:
Objective image quality - signal-to-noise and contrast-to-noise ratio | Measurement for each scan is performed within 1 month after the scan.
  The objective image quality parameters consist of signal-to-noise ratio (SNR) and contrast-to-noise ratio (CNR). SNR is calculated by dividing the attenuation of the liver parenchyma by the corresponding standard deviation (SD) of the attenuation. The attenuation of the left erector spinae muscle is measured at the level of the liver to calculate CNR using the following established formula: liver segment attenuation minus intramuscular attenuation, divided by the SD of the intramuscular attenuation. For both a higher number indicated a better image quality. The outcome should not be significantly different between groups.
Subjective image quality - assessed with a 5-point Likert scale | Measurement for each scan is performed within 1 month after the scan.
  Two experienced radiologists will assess the subjective image quality in consensus, while being blinded for the protocol used. A 5-point Likert scale is used, in which 1= excellent; 2= good; 3 = moderate; 4 = poor; 5 = very poor. So a higher number is a worse outcome. The scale does not have a particular name.
Radiation dose | Measurement for each scan is performed within 1 month after the scan.
  The mean effective mAs (± SD), mean CTDIvol (mGy) (± SD) and the Mean DLP (mGy*cm) (± SD) are visible on screen and reported, to compare the difference in radiation dose between groups. A higher number means a higher radiation dose and is therefore a worse outcome.
Weight | Directly prior to the scan it is measured and data is collected within one month after the scan.
  Patients weight (in kg) is assessed by using a weighting scale
Height (in m) | Directly prior to the scan it is measured and data is collected within one month after the scan.
  Patients height is asked
Contrast media volume | Data is retrieved from the system within 1 month after the scan.
  A dedicated data acquisition program (Certega Informatics Solution; Bayer) continuously monitors and collects all injection parameters (eg, total amount of CM [milliliter] and peak flow rate [milliliter per seconds]). A higher number means a higher radiation dose and is therefore a worse outcome. And results are compared between groups.
Needle size | Data is retrieved from the system within 1 month after the scan. It is finished when all patients are scanned.
  A dedicated data acquisition program (Certega Informatics Solution; Bayer) continuously monitors and collects all injection parameters, among which needle size is one of the parameters. A smaller gauge of the needle could possibly mean that the desired flow rate is not possible. In general it is expected that the needle size used is not significantly different between groups.
Needle placement | Data is retrieved from the system within 1 month after the scan.
  A dedicated data acquisition program (Certega Informatics Solution; Bayer) continuously monitors and collects all injection parameters, among which needle placement is one of the parameters. In general it is expected that the needle placement is not significantly different between groups.
BMI | Calculated after the scan, within 1 month after the scan.
  Weight and height will be combined to report BMI in kg/m^2
Sex | Collected before the scan by the technician and retrieved from the system within 1 month after the scan.
  Is collected
Age | Collected before the scan by the technician and retrieved from the system within 1 month after the scan.
  Is collected
Scan indication | Collected before the scan by the technician and retrieved from the system within 1 month after the scan.
  Is collected
Flow rate | Data is retrieved from the system within 1 month after the scan.
  A dedicated data acquisition program (Certega Informatics Solution; Bayer) continuously monitors and collects peak flow rate [milliliter per seconds]).
Concentration of the contrast media | Data is retrieved from the system within 1 month after the scan.
  All patients receive the identical contrast media concentration as used in daily clinical routine; 300 mg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Wildberger, Professor, Principal Investigator — Maastricht University Medical Center
Locations (1):
- MUMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.